CLINICAL TRIAL: NCT00463944
Title: Assessment of an Electronic Voting System Within the Tutorial Setting. A Randomised Controlled Trial
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Other Study IDs: 1
Record Dates: First submitted 2005-06-30; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2005-06

CONDITIONS: Healthy
Keywords: Electronic voting system

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Effect of an electronic voting system

SUMMARY:
A study of an electronic voting system as a learning aid during tutorials

DETAILED DESCRIPTION:
A study of an electronic voting system as a learning aid during tutorials. This study was undertaken with clinical students over a one year period of observation

ELIGIBILITY:
Inclusion Criteria:

* All fourth year students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 2001-01; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Peter Devitt, Principal Investigator — University of Adelaide
Locations (1):
- University of Adelaide, Adelaide, South Australia, Australia